CLINICAL TRIAL: NCT02075021
Title: Phase I/II Trial of the Combination of Lenalidomide (Revlimid) and Nab-paclitaxel (Abraxane) in the Treatment of Relapsed/Refractory Multiple Myeloma
Acronym: rev/abraxane
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI left the institution
Sponsor: NYU Langone Health (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-02519
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2017-09-05 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Relapsed or Refractory Multiple Myeloma
Keywords: relapsed; refractory; multiple myeloma; revlimid; lenalidomide; abraxane; n-paclitaxel
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Lenalidomide; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- lenalidomide and nab-paclitaxel (Experimental): 100 mg/m^2 of Abraxane weekly for 3 weeks and 10 mg Revlimid daily for 21 days, with a dose escalation for Revlimid to 15 mg and to 25 mg. One cycle is 4 weeks. Dose de-escalations will also be performed for both drugs as necessary. Patients will be treated until disease progression.
  Interventions: Drug: Lenalidomide; Drug: nab-paclitaxel

INTERVENTIONS:
Drug: Lenalidomide
  Other Names: Revlimid
Drug: nab-paclitaxel
  Other Names: Abraxane

SUMMARY:
The investigators will perform a phase I/II trial of Revlimid daily for 21 days and Abraxane weekly for 3 weeks. Accrual will be on standard cohorts of 3 patients. Once the maximum toxicity dose (MTD) is reached, the level below will be expanded to 25 patients for a pilot phase II trial. All treatments will be performed until progression. Assessments will be made at least at the 2, 4 and 6 month timepoints and monthly thereafter until progression.

The purpose of this research study is to determine how much of the combination of Revlimid and Abraxane can be given safely and how well they work together against the cancer.

Currently, this trial is in the phase 1 stage.

DETAILED DESCRIPTION:
Revlimid is an important imid based therapy of myeloma. However patients will still relapse after this drug and then have limited options. Abraxane has shown efficacy in a number of cancers, putatively through intratumor concentration by SPARC (secreted protein acidic and rich in cysteine). (Taxanes have shown a modest activity in myeloma. Interestingly, Revlimid can upregulate the levels of SPARC. Thus, investigators will test the toxicity and efficacy of a combination of Revlimid and Abraxane in relapsed/refractory myeloma.

Investigators will perform a phase I/II trial of Revlimid daily for 21 days and Abraxane weekly for 3 weeks in patients who have failed Revlimid but have adequate blood counts and renal function and minimal neuropathy. For study purposes, 1 cycle is considered to be 4 weeks (20 days). Subjects will get Abraxane for three weeks and will be off of this treatment for 1 week. There are 10 visits per cycle. Accrual will be on standard 3 patient cohorts. Once the maximum tolerated dose is reached, the level below will be expanded to 25 patients for a pilot phase II trial. All treatments will be performed until progression. Assessments will be made at least at the 2, 4, and 6 month timepoints and monthly thereafter until progression.

Since both drugs can cause myelosuppression, investigators will start with doses below their standard doses as single agents. Investigators will use 100 mg/m2 of Abraxane weekly for 3 weeks and 10 mg Revlimid daily for 21 days, with a dose escalation for Revlimid to 15 mg and to 25 mg. Dose de-escalations will also be performed for both drugs as necessary. Investigators will explore whether SPARC (secreted protein acidic and rich in cysteine) expression is altered by flow cytometry and immunohistochemistry.

ELIGIBILITY:
Inclusion Criteria:

* Patients with relapsed/refractory multiple myeloma based on standard criteria
* Renal function assessed by calculated creatinine clearance as follows
* Phase I subjects must have calculated creatinine clearance >=30ml/min by Cockcroft-Gault formula.
* Phase II subjects must have calculated creatinine clearance >=30ml/min by Cockcroft-Gault formula.
* Progressed (>25% increase in evaluable disease) or non response on Revlimid or within 60 days of stopping Revlimid
* > 1 prior regimen
* Total bilirubin <=1.5 x Upper limit of normal (ULN)
* AST (aspartate aminotransferase) or serum glutamic-oxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT) or serum glutamic-pyruvic transaminase (SGPT) <=3 x ULN.
* All study participants must be registered into the mandatory Revlimid REMS® program, and be willing and able to comply with the requirements of Revlimid REMS®.
* Females of childbearing potential must have a negative serum or urine pregnancy test with a sensitivity of at least 50 mIU/mL (milli-International unit/milliliter) within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days as required by Revlimid REMS) and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide.
* Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA (acetylsalicylic acid) may use warfarin or low molecular weight heparin).
* With < or = grade 2 neuropathy
* Karnofsky performance status ≥ 50
* Patients treated with local radiotherapy with or without a brief (2 weeks or less) exposure to steroids are eligible. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed
* Meets the following pretreatment laboratory criteria at Baseline (Day 1 of Cycle 1, before study drug administration)

  1. Platelet count ≥ 75 x 10^3/uL (upper limit) .
  2. Hemoglobin ≥ 8.0 g/dL (grams/deciliter)
  3. Absolute neutrophil count ≥ 1.0 x 10^3/uL
* Age 18 years or older

Exclusion Criteria:

* > grade 2 neuropathy
* > Cr (complete response) 2.5
* LFTs (liver function test) > 2x nl (normal limit)
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG (electrocardiogram) abnormality at screening must be documented by the investigator as not medically relevant.
* Known hypersensitivity to thalidomide or Revlimid (if applicable).
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis B virus vaccine are eligible.
* Female subject is pregnant or lactating. Confirmation that the subject is not pregnant must be established by a negative serum -human chorionic gonadotropin (hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for postmenopausal or surgically sterilized women.
* Female patients who are lactating or have a positive serum pregnancy test during the screening period, or a positive urine pregnancy test on Day 1 before first dose of study drug, if applicable.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Radiation therapy within 3 weeks before randomization. Enrollment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 3 weeks have elapsed since the last date of therapy.
* POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes)
* Plasma cell leukemia
* Receiving steroids daily for other medical conditions, e.g., asthma, systemic lupus erythematosis, rheumatoid arthritis
* Infection not controlled by antibiotics
* HIV infection. Patients should provide consent for HIV testing according to the institution's standard practice
* Known active hepatitis B or C

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-03; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amitabha Mazumder, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU School of Medicine, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Confirmed diagnosis of relapsed/refractory multiple myeloma.
Groups:
- Lenalidomide and Nab-paclitaxel: 100 mg/m^2 of Abraxane weekly for 3 weeks and 10 mg Revlimid daily for 21 days, with a dose escalation for Revlimid to 15 mg and to 25 mg. One cycle is 4 weeks. Dose de-escalations will also be performed for both drugs as necessary. Patients will be treated until disease progression.
  Lenalidomide
  nab-paclitaxel
Period: Overall Study
Arm/Group | Lenalidomide and Nab-paclitaxel
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 3 Subjects accrued and completed follow up. Data was not analyzed because PI left institution.
Arm/Group | Lenalidomide and Nab-paclitaxel
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (Phase I)
Description: Dose limiting toxicity will be accessed based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: 4 weeks
Population: Results were not analyzed due to lack of sufficient data. PI left the institution.
Arm/Group | Lenalidomide and Nab-paclitaxel
Number analyzed (Participants) | 0

2. Secondary Outcome: the Number of Patients Who Achieve Complete Response (CR) or Partial Response (PR) (Phase II)
Description: The response will be determined using the International Uniform Response Criteria for Multiple Myeloma.
Time Frame: up to 2 years
Population: Results were not analyzed due to lack of sufficient data. PI left the institution.
Arm/Group | Lenalidomide and Nab-paclitaxel
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Lenalidomide and Nab-paclitaxel
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No